CLINICAL TRIAL: NCT05219513
Title: An Open-Label, Phase 1 Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of RO7443904 in Combination With Glofitamab in Participants With Relapsed/Refractory B-Cell Non-Hodgkin's Lymphoma
Brief Title: A Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Efficacy of RO7443904 in Combination With Glofitamab in Participants With Relapsed/Refractory B-Cell Non-Hodgkin's Lymphoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was terminated due to sponsor portfolio re-alignment.
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BP43131
Record Dates: First submitted 2021-11-23; First posted 2022-02-02 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Lymphoma, Non-Hodgkin
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — glofitamab; obinutuzumab; tocilizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Parts I-III: Dose-escalation of RO7443904 (Experimental): The dose-escalation of RO7443904 and glofitamab will take place every three weeks (Q3W) with obinutuzumab pre-treatment.
  Interventions: Drug: RO7443904; Drug: Glofitamab; Drug: Obinutuzumab; Drug: Tocilizumab
- Part IV: Dose-expansion of RO7443904 (Experimental): Part IV of this study will evaluate selected dose levels of RO7443904 in combination with glofitamab from Parts I-III in a Q3W regimen with obinutuzumab pre-treatment.
  Interventions: Drug: RO7443904; Drug: Glofitamab; Drug: Tocilizumab

INTERVENTIONS:
Drug: RO7443904 — RO7443904 will be administered by subcutaneous (SC) or IV infusion on Cycle (C) 1 Day (D) 10, C2D3, and C2D8. From C3 onward, RO7443904 will be given every 3 weeks (Q3W), for up to 12 cycles (C = 21 days).
Drug: Glofitamab — Glofitamab will be administered through IV infusion starting with step-up dosing (2.5 mg/10 mg/30 mg) on C1D1, C1D8, and C2D1. Starting in Cycle 3, glofitamab will be given in 30 mg doses every three weeks (Q3W) with RO7443904, for up to 12 cycles (Cycle = 21 days).
  Other Names: RO7082859
Drug: Obinutuzumab — Obinutuzumab will be administered once through IV infusion, at a 1 g dose in Cycle 1, on either Day -7, -4, or -3 (C1D-7, C1D-4, C1D-3).
  Arms: Parts I-III: Dose-escalation of RO7443904
Drug: Tocilizumab — Tocilizumab will be administered as necessary to treat cytokine release syndrome (CRS).
  Other Names: Actemra

SUMMARY:
This is a first-in human, open-label, Phase 1 dose-escalation study in order to determine the maximum tolerated dose (MTD) and/or recommended Phase 2 dose (RP2D) for intravenous (IV) and/or subcutaneous (SC) dosing schemes of this combination treatment, and to evaluate the safety, tolerability, pharmacokinetics, and preliminary anti-tumor activity of this combination treatment in participants with relapsed/refractory B-cell non Hodgkin lymphoma (r/r NHL).

ELIGIBILITY:
Inclusion Criteria:

* Body weight >=40 kg
* Histologically confirmed hematological malignancy that is expected to express CD19 and CD20 and with clinical evidence of treatment need; 2) relapse after or failure to respond to at least two prior treatment regimens; and 3) no other available treatment options that are known to provide clinical benefit
* Must have at least one measurable target lesion (>=1.5 cm) in its largest dimension by computed tomography (CT) scan
* Able and willing to provide a fresh tumor biopsy from a safely accessible site, per Investigator's determination
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Life expectancy of >=12 weeks
* Adequate liver, hematological and renal function
* Negative serologic or polymerase chain reaction (PCR) test results for acute or chronic hepatitis B virus (HBV) infection
* Negative test results for hepatitis C virus (HCV) and HIV
* A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies: 1) Women of non-childbearing potential 2) Women of childbearing potential (WOCBP), who, agree to remain abstinent (refrain from heterosexual intercourse) or use of one highly effective contraceptive method during the treatment period and for at least 18 months after obinutuzumab or 5 months after the final dose of RO7443904, 2 months after final dose of glofitamab or 3 months after the final dose of tocilizumab
* Male participants must remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures such as a condom plus an additional contraceptive method with a partner who is a WOCBP during the treatment period and for at least 3 months after obinutuzumab, 5 months after the final dose of RO7443904, 2 months after the final dose of glofitamab or 2 months after the final dose of tocilizumab, whichever is longer

Exclusion Criteria:

* Circulating lymphoma cells, defined by out-of-range (high) absolute lymphocyte count (ALC) or the presence of abnormal cells in the peripheral blood signifying circulating lymphoma cells
* Participants with known acute bacterial, viral, or fungal infection 72 hours prior to glofitamab infusion
* Participants with known active infection or reactivation of a latent infection
* Pregnant, breastfeeding, or intending to become pregnant during the study
* Prior treatment with systemic immunotherapeutic agents
* History of treatment-emergent, immune-related adverse events (AEs) associated with prior immunotherapeutic agents
* Persistent AEs from prior anti-cancer therapy Grade >=1
* Treatment with standard radiotherapy, any chemotherapeutic agent, or treatment with any other investigational or approved anti-cancer agent
* Prior solid organ transplantation
* Prior allogeneic stem cell transplant (SCT)
* Autologous SCT within 100 days prior to obinutuzumab infusion
* Autoimmune disease in active phase or exacerbation/flare within at least 6 months of enrollment
* History of immune deficiency disease that increases the risk of infection
* History of contraindication and/or severe allergic or anaphylactic reactions to monoclonal antibody therapy and/or prophylactic drugs used for cytokine release syndrome (CRS) and tumor lysis syndrome (TLS)
* History of confirmed progressive multifocal leukoencephalopathy
* Current or past history of central nervous system (CNS) lymphoma or CNS disease
* Evidence of significant, uncontrolled concomitant diseases that could affect compliance with the protocol or interpretation of results
* Major surgery or significant traumatic injury <28 days prior to the GpT infusion or anticipation of the need for major surgery during study treatment
* Participants with another invasive malignancy in the last 2 years
* Significant cardiovascular disease
* Administration of a live, attenuated vaccine within 4 weeks before GpT infusion or anticipation that such a live attenuated vaccine will be required during the study
* Received systemic immunosuppressive medications for reasons other than anticancer therapy within the last 6 months of enrollment with the exception of corticosteroid treatment <= 25 mg/day prednisone or equivalent
* History of illicit drug or alcohol abuse within 12 months prior to screening, in the Investigator's judgment
* Any other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that would contraindicate the use of an investigational drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2022-02-18 (Actual); Primary Completion 2024-07-17 (Actual); Study Completion 2024-07-17 (Actual)

PRIMARY OUTCOMES:
Nature and frequency of dose-limiting toxicities (DLTs) | From 3 weeks (21 days) from the first administration of RO7443904 (Cycle 2 Day 8) to 1 week after the second administration of RO7443904 (Cycle 3 Day 8)
Incidence, nature, and severity of AEs | Up to 4 weeks after the last study treatment dose
  graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v5.0 and for cytokine-release syndrome (CRS) and neurotoxicity (immune effector cell-associated neurotoxicity syndrome; ICANS) according to the American Society for Transplantation and Cellular Therapy (ASTCT) consensus grading

SECONDARY OUTCOMES:
Maximum concentration (Cmax) of RO7443904 | Up to 9 months
Area under the curve (AUC) of RO7443904 | Up to 9 months
Clearance (CL) of RO7443904 | Up to 9 months
Volume of distribution (Vd) of RO7443904 | Up to 9 months
Half-life (t1/2) of RO7443904 | Up to 9 months
Percentage of Participants with RO7443904 anti-drug antibodies (ADAs) during the study relative to the prevalence of ADA at baseline | Up to 9 months
Time to maximum concentration (Tmax) of RO7443904 | Up to 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (9):
- United States (3):
  - MSKCC, New York, New York
  - Cleveland Clinic Foundation; Hematology and Oncology, Cleveland, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
- Peter MacCallum Cancer Centre; Department of Haematology, Melbourne, Victoria, Australia
- Rigshospitalet; Hæmatologisk Klinik, Klinisk Afprøvnings Team KAT, København Ø, Denmark
- CHRU Lille - Hôpital Claude Huriez; Service des Maladies du Sang, Lille, France
- Italy (2):
  - ASST PAPA GIOVANNI XXIII; Ematologia, Bergamo, Lombardy
  - Istituto Clinico Humanitas;U.O. Oncologia Medica Ed Ematologia, Rozzano, Lombardy
- Leicester Royal Infirmary; Dept of Haematology, Leicester, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.clinicalstudydatarequest.com). Further details on Roche's criteria for eligible studies are available here (https://clinicalstudydatarequest.com/Study-Sponsors/Study-Sponsors-Roche.aspx). For further details on Roche's Global Policy on Sharing of Clinical Study Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm)

REFERENCES:
- [Derived] Sam J, Hofer T, Kuettel C, Claus C, Thom J, Herter S, Georges G, Korfi K, Lechmann M, Eigenmann MJ, Marbach D, Jamois C, Lechner K, Krishnan SM, Gaillard B, Marinho J, Kronenberg S, Kunz L, Wilson S, Briner S, Gebhardt S, Varol A, Appelt B, Nicolini V, Speziale D, Bez M, Bommer E, Eckmann J, Hage C, Limani F, Jenni S, Schoenle A, Le Clech M, Vallier JP, Colombetti S, Bacac M, Gasser S, Klein C, Umana P. CD19-CD28: an affinity-optimized CD28 agonist for combination with glofitamab (CD20-TCB) as off-the-shelf immunotherapy. Blood. 2024 May 23;143(21):2152-2165. doi: 10.1182/blood.2023023381. PMID 38437725